CLINICAL TRIAL: NCT00964483
Title: Translating the Dietary Approaches to Stop Hypertension (DASH)Diet Into an Urban, African-American Community in Winston-Salem, North Carolina
Brief Title: Translating Dietary Trials Into the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Gramercy Research Group (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R21HL091303-02 (NIH); 5R21HL091303-02 (NIH)
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DASH materials (Experimental): Participant randomized to a 12-week, group-based lifestyle intervention using modified DASH materials and intervention delivery approaches to help them adopt the DASH diet. Intervention content will be designed to provide participants with the knowledge and skills to adopt the DASH eating pattern, specifically to increase fruit, vegetable, and low-fat dairy intake, and to decrease saturated fats and sodium.
  Interventions: Behavioral: DASH diet
- Delayed intervention (Active Comparator): The intervention participants will receive an NHLBI brochure entitled "Your Guide to Lowering Blood Pressure." They will then receive the modified DASH materials and the intervention at the end of the study, following the intervention group's completion of the study.
  Interventions: Behavioral: DASH diet; Behavioral: Delayed Intervention

INTERVENTIONS:
Behavioral: DASH diet — The intervention will consist of a 12-week pilot trial in which participants will be given intervention materials tailored to their community, focusing on DASH. Intervention content will be designed to provide participants with the knowledge and skills to adopt the DASH eating pattern, specifically to increase fruit, vegetable, and low-fat dairy intake, and to decrease saturated fats and sodium. They will follow this diet for 12 weeks.
Behavioral: Delayed Intervention — The participants will receive a guide written by NHLBI entitled, "Your Guide to Lowering Blood Pressure."
  Arms: Delayed intervention

SUMMARY:
A diet that is rich in fruits, vegetables, and low fat dairy foods is known to lower blood pressure in adults. This research project seeks to promote the adoption of the Dietary Approaches to Stop Hypertension(DASH)eating pattern by African American adults with hypertension or prehypertension living in a lower income minority community. The randomized trial phase of this project will test a group-based intervention using materials adopted from prior studies and tailored to the community of interest.

DETAILED DESCRIPTION:
Hypertension (HTN) is a prevalent risk factor for cardiovascular, cerebrovascular, and renal disease, and disproportionately affects African Americans (AA). Although HTN awareness and treatment rates among AA are similar to, or exceed non-Hispanic whites, control of HTN among AAs remains inadequate. Randomized clinical trials have demonstrated the effectiveness of lifestyle measures in lowering BP, including the Dietary Approaches to Stop Hypertension (DASH) diet, which lowers systolic BP 6-14 mmHg. DASH calls for increased consumption of fruits, vegetables, and low fat dairy, and decreased saturated fat and sodium intake. There is limited evidence that DASH has been widely adopted by the public and AA from lower income communities may be less able to adopt DASH as currently disseminated due to barriers related to income, education, attitudes about foods, health beliefs, and neighborhood availability of healthier foods. We propose to utilize quantitative and qualitative research techniques (including focus groups and surveys) to assess environmental, intra-personal, interpersonal and cultural factors that could affect the translation of the DASH diet in a low-income AA community, then utilize the knowledge gathered to adapt existing intervention strategies and tools. These will provide the materials for a randomized three month pilot lifestyle intervention implementing the DASH diet. The 40 participants will be aged 21+ and have pre-HTN or HTN with blood pressure between 120-150/80-95 mmHg on 0,1 or 2 antihypertensive agents, and will be AA residents of two zip codes in Winston-Salem (a lower-income area whose population is significantly minority).

ELIGIBILITY:
Inclusion Criteria:

* Being African American
* Age 21 years or older
* Residing in zip code 27105 or 27101
* Formal education less than 4-year college degree
* Blood pressure between 120/80 mmHg and 150/95 mmHg, inclusive (patients on BP lowering drugs eligible if BP is in above range)
* Willing to provide informed consent
* Able to participate in English

Exclusion Criteria:

* Clinical history of congestive heart failure
* Clinical history of diabetes, or newly diagnosed diabetes at screening
* Clinical history of renal insufficiency (Stage 3 or higher chronic kidney disease)
* BMI less than or equal to 18.5 kg/m2 or greater than or equal to 45.0 kg/m2
* Pregnancy
* Non-English speaker

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Dietary change from baseline. | Three Months

SECONDARY OUTCOMES:
Participation | three months
Blood pressure | three months

CONTACTS AND LOCATIONS:
Overall Officials: Alain G Bertoni, MD, MPH, Principal Investigator — Wake Forest University Health Sciences; Melicia C Whitt-Glover, PhD, Principal Investigator — Gramercy Research Group
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided